CLINICAL TRIAL: NCT04828096
Title: Retention With Three Different Bonded Retainers: a Multicenter, Randomized Controlled Trial With 5-year Follow-up
Brief Title: Retention With Three Different Bonded Retainers a Multicenter, Randomized Controlled Trial With 5-year Follow-up
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Farhan Bazargani, DDS, PhD, Associate professor, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-04104
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Dental Malocclusion; Stability
Keywords: Orthodontic retention, Stability, Long-term
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Penta-one retainer (Active Comparator): Penta-one retainer is one wire that is been in use for many years. Penta-one retainer is to be bonded on the lower anterior 6 teeth (canine-to-canine)- Half of the retainers are going to be bonded with sandblasted enamel and half without.
  Interventions: Other: Orthodontic retention
- Ortho-FlexTech retainer (Experimental): Ortho-Flextech chain wire is relatively new in the market and needs to be evaluated. Ortho-Flextech retainer is to be bonded on the lower anterior 6 teeth (canine-to-canine)- Half of the retianers are going to be bonded with sandblasted enamel and half without.
  Interventions: Other: Orthodontic retention
- Memotain retainer (Experimental): Memotain wire is relatively new in the market. It requires digital scanning and the technique is said to be very exact. Memotain retainer is to be bonded on the lower anterior 6 teeth (canine-to-canine)- Half of the retianers are going to be bonded with sandblasted enamel and half without.
  Interventions: Other: Orthodontic retention

INTERVENTIONS:
Other: Orthodontic retention — The stability of the mandibular anterior teeth after two resp. 5 years of retention

SUMMARY:
One of major challenges in orthodontics is to inhibit relapse and ensure stability of treatment outcomes. Retention is the phase of orthodontic treatment that attempts to keep teeth in the corrected position after correction with orthodontic braces. Without retention there is a tendency for the teeth to return to their initial position (1). Retention is usually necessary to overcome the elastic recoil of the periodontal supporting fibers and to allow remodeling of the alveolar bone. The bonded orthodontic lingual retainer constructed from composite and orthodontic wires provides an esthetic and efficient system for maintained retention and has been shown to be an effective means of retaining aligned anterior teeth in the post treatment position in the long term. This has been in popular use as a method of retention since the late 1970s (2).

The traditional retainers, which are still in use, are multi-strand stainless steel retainers such as Penta-one® 0.0215 (Masel Orthodontics, Carlsbad, CA, USA). The main problem with multistrand stainless steel retainers is their high rate of failure. Clinical studies indicate that 5% to 37% of mandibular retainers fail during retention in some form, either bond failure or wire breakage (3-5). Reliance Orthodontic Products, Inc. (Itasca, IL, USA) recently introduced a bonded retainer system (Ortho-Flextech™ chain). This retainer's bonding is claimed to be quick and easy by reducing chairside time and eliminating laboratory costs (6). One other recently introduced retainer is Memotain™ (CA-Digital in Mettmann, Germany). Memotain is a CAD/CAM fabricated lingual retainer made of 0.014 X 0.014-inch rectangular nickel-titanium. The wire is highly flexible and custom cut to precisely adapt to the patient's lingual tooth anatomy. According to manufacturer, Memotain offers numerous perceived advantages to traditional multistranded lingual wires, including no need for wire measuring or bending, individually optimized placement, greater accuracy of fit, tighter interproximal adaptation, less tongue irritation, better durability, and resistance to microbial colonization (6). However, randomized clinical trials are necessary to determine whether these advantages are substantiated with scientific data.

A recent review by the Cochrane group concluded that to date there is insufficient evidence to single out any particular retention strategy as the preferred method: it was recommended that future studies should include true randomization, reporting of dropouts, adequate sample size calculation, and a minimum follow-up period of 3 months (8). Thus, the aims of this multicenter, randomised controlled trial are:

* To compare and evaluate the effectiveness and failure rate of Penta-one multistrand, Ortho-Flextech and Memotain retainers with each other
* To compare the possible complications between the three retainers over time
* To establish the cost-effectiveness of the three retainers
* To evaluate the effectiveness of sandblasting in the retention of the wires

DETAILED DESCRIPTION:
Trial design This study is a 3-arm parallel-group, randomized controlled trial with a 1:1 allocation ratio.

Participants, eligibility criteria, and setting

Participants are to be recruited at the Postgraduate Dental Education Center, Department of Orthodontics, in Örebro, Henrikson Orthodontics, in Malmö and Universitat Internacional de Catalunya, Department of Orthodontics, in Barcelona.

The following inclusion criteria is to be applied:

* Patients requiring mandibular lingual fixed canine-to-canine retainer after undergoing orthodontic treatment with fixed appliances
* Sound enamel on the lingual surface
* Calculus-free lingual surface in the lower anterior segment

Interventions

After informed consent is obtained, the patients are going to be randomized into three groups:

Group 1: Penta-One 0.0215 inch multistranded wire

Group 2: Ortho-FlexTech stainless steel chain

Group 3: Memotain wire

Procedures For all groups the time required for taking impressions and bonding of retainers is taken by a digital timer.

Patients allocated to Group 1:

After taking impressions and when the working models are cast in hard stone, all retainers (0.0215-inch multistranded Penta-one wire) are going to be contoured by dental technicians at each center.

All retainers in the study are to be bonded using the following sequence of construction.

* The fixed appliance is debonded, and the teeth are to be thoroughly cleaned and polished using oil-free pumice.
* After adequate moisture control using dental cotton rolls in the anterior segment, parotis dental rolls in the lateral segments, and saliva ejector, the lingual surfaces are to be sandblasted in half of the group (according to the randomization list)
* Lingual surfaces are etched with Ultra-Etch 35% phosphoric acid gel (Ultradent Products Inc, City, Utah), for 30 seconds and thoroughly rinsed and dried.
* A thin layer of primer Ortho Solo® (Ormco, Orange, CA, USA) applies.
* Retainer holds in place with dental floss and the fit is checked.
* Adequate amounts of composite Tetric Evo-Flow (Ivoclar Vivadent, Schaan, Liechtenstein) is applied to the lingual surfaces of the six anterior teeth over the retainer, ensuring maximum coverage of the wire surface. The composite pads are light cured, both incisally and cervically, for 20 seconds per tooth.

Patients allocated to Group 2:

* The fixed appliance is debonded, and the teeth are to be thoroughly cleaned and polished using oil-free pumice.
* After adequate moisture control using dental cotton rolls in the anterior segment, parotis dental rolls in the lateral segments, and saliva ejector, the lingual surfaces are to be sandblasted in half of the group (according to the randomization list)
* Lingual surfaces are etched with Ultra-Etch 35% phosphoric acid gel (Ultradent Products Inc, City, Utah), for 30 seconds and thoroughly rinsed and dried.
* A thin layer of primer Ortho Solo® (Ormco, Orange, CA, USA) applies.
* Small amounts of composite Tetric Evo-Flow (Ivoclar Vivadent, Schaan, Liechtenstein) were applied to the lingual surfaces of the six anterior teeth.
* Ortho-FlexTech chain is cut at chairside in desired length and hold in place with dental floss and the fit is checked.
* Small amounts of composite Tetric Evo-Flow (Ivoclar Vivadent, Schaan, Liechtenstein) is applied to the lingual surfaces of the six anterior teeth over the retainer, ensuring maximum coverage of the wire surface. The composite pads are light cured, both incisally and cervically, for 20 seconds per tooth. Additional composite applies to cover the whole mesial-deistal surface of each tooth making sure not to cover the approximal surfaces. Then light cured for another 20 second per tooth.

Patients allocated to Group 3:

* After digital scanning of the anterior lower six teeth, the Memotain in ordered online.
* The fixed appliance is debonded, and the teeth are to be thoroughly cleaned and polished using oil-free pumice.
* After adequate moisture control using dental cotton rolls in the anterior segment, parotis dental rolls in the lateral segments, and saliva ejector, the lingual surfaces are to be sandblasted in half of the group (according to the randomization list)
* Lingual surfaces are etched with Ultra-Etch 35% phosphoric acid gel (Ultradent Products Inc, City, Utah), for 30 seconds and thoroughly rinsed and dried.
* A thin layer of primer Ortho Solo® (Ormco, Orange, CA, USA) applies.
* Memotain puts into placed using the positioning jig to ensure precise placement.
* Adequate amounts of composite Tetric Evo-Flow (Ivoclar Vivadent, Schaan, Liechtenstein) are applied to the lingual surfaces of the canines initially and after removing the positioning jig on the remaining four anterior teeth, ensuring maximum coverage of the wire surface. The composite pads are light cured, both incisally and cervically, for 20 seconds per tooth.

Follow-ups During the visit to the clinics all groups are to take impressions with digital scanning of the upper and the lower dentition and intraoral photographs from the dentition at baseline (directly after debond) T0, 6 months after debond (T1), one year (T2) two years (T3) and five years (T4) after debond.

The digital study models will be assessed for identifying possible side effects and deviation of individual tooth positions. For this purpose Little's Irregularity Index (LII) (9) for tooth contact displacement will be used. Patients' records will be reviewed to assess the first debond or breakage of the retainers during the observation periods.

To determine the cost-effectiveness, the overall cost of the retainers including manufacturing, time for impressions and bonding will be calculated and compared.

Failure of a retainer can occur as a result of debonding, fracture, debonding and fracture, or retainer loss. Information on the site of failure e.g. single tooth bond failure, enamel/adhesive failure, or adhesive wire failure is to be recorded in the patients' records.

Only ﬁrst failures are to be counted and failure location (which tooth) is to be noted. In addition, multiple failure sites in one retainer are going to be counted as one failure. Furthermore, failure is considered when there was debonding, fracture, debonding and fracture, or retainer loss.

Outcomes The primary outcome is failure rate/breakage of the retainers during the observation period.

Secondary outcome include, complications (such as BoP, calculus, caries, gingivitis), costs and the effect of micro-etching (sand blasting) on the failure rate.

Sample size estimation The calculated sample size for each group is based on a significance level of 0.05 and 90 per cent power to detect a clinically meaningful difference of 15 per cent failure rate between the groups. The sample size calculation indicated that 97 patients would be required in each group. To compensate for dropouts, we decided to include at least 108 patients in each group (an addition of 10 per cent per group) and a total of 324 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring mandibular lingual fixed canine-to-canine retainer after undergoing orthodontic treatment with fixed appliances
* Sound enamel on the lingual surface
* Calculus-free lingual surface in the lower anterior segment

Exclusion Criteria:

-

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 324 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Failure rate | 2-year follow-up
  Failure rate/breakage of the retainers during the observation periods
Failure rate | 5-year follow-up
  Failure rate/breakage of the retainers during the observation periods

SECONDARY OUTCOMES:
Complications | 2-year follow-up
  Incidence of complications (if any) such as retraction of gingival tissue
Cost-effectiveness | 2-year follow-up
  Cost-effectiveness analysis
Effect of micro-etching | 2-year follow-up
  Effect of sandblasting on bonding strength and failure rate is to be evaluated
Complications | 5-year follow-up
  Incidence of complications (if any) such as retraction of gingival tissue
Cost-effectiveness | 5-year follow-up
  Cost-effectiveness analysis
Effect of micro-etching | 5 -year follow-up
  Effect of sandblasting on bonding strength and failure rate is to be evaluated

CONTACTS AND LOCATIONS:
Locations (2):
- Universitat Internacional de Catalunya, Department of Orthodontics, Barcelona, Catalonia, Spain
- Postgraduate Dental Education Center, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.